CLINICAL TRIAL: NCT00176514
Title: A Pilot Trial to Assess the Effects of Green Tea in the Prevention of Therapy-Induced Mucositis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Susan Goodin, PhD, UMDNJ/CINJ
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3074; 060001 (Other: CINJ)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Mucositis
Keywords: mucositis
MeSH Terms: conditions — Mucositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Administration of the antineoplastic

SUMMARY:
This is a clinical research study that is designed to determine if there is a potential benefit of green tea to help treat and prevent therapy induced mucositis, which is mouth sores caused by chemotherapy.

DETAILED DESCRIPTION:
The overall objective of this study is to assess the effect of green tea on reducing the incidence or severity of chemotherapy (with or without radiotherapy) induced mucositis in patients receiving standard therapy that will produce a very high likelihood of oral, esophageal, or gastrointestinal mucositis (e.g. high dose chemotherapy with stem cell reconstitution in patients with multiple myeloma; concurrent 5-FU/ cisplatin and radiotherapy to the head and neck area; patients receiving paclitaxel).

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed diagnosis of cancer for which standard chemotherapy will produce a very high likelihood of oral, esophageal or gastrointestinal mucositis (e.g. high dose chemotherapy with stem cell reconstitution in patients with multiple myeloma; concurrent 5-FU/ cisplatin and radiotherapy to the head and neck area; patients receiving paclitaxel). Patients receiving concurrent chemotherapy/radiation therapy for lung or gastrointestinal cancer are eligible.

If not receiving a highly mucosally toxic regimen, have had Grade 2 mucositis on the prior cycle of chemotherapy Have no evidence of active infection in the oral cavity such as thrush, HSV, or aphthous ulcers.

Patients must be free of known infectious stomatitis or systemic infection (culture not required). If unclear that the patient has infectious stomatitis, cultures may be obtained and the patient entered on study.

Must be free of Grade 3 or 4 vomiting. Have no contraindication for buccal scrapings. Not be a frequent (>3 cups per day) tea drinker Must be able to speak English.

Exclusion Criteria:

Xerostomia Use of any investigational agent (not FDA approved) Current use of, allopurinol, prostaglandin inhibitors, sulcralfate, vitamin E or antioxidant supplements during the course of this study.

Patients receiving an anesthetic "cocktail" regimen or other topical anesthetics.

Patients with existing oral lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37
Dates: Start 2000-07; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Assess the effect of tea on reducing the incidence or severity of chemotherapy induced mucositis

SECONDARY OUTCOMES:
Correlate the levels of tea polyphenols in buccal cells and in saliva with the effect of tea on the change in incidence or severity of treatment induced mucositis.
Correlate the analyses of proliferation index, cyclooxygenase, and prostagladin E- 2 with the change in incidence or severity of chemotherapy induced mucositis.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Goodin, PharmD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Cancer Institute of New Jersey, New Brunswick, New Jersey, United States